CLINICAL TRIAL: NCT00486343
Title: A Randomized, Double-Blind, Placebo Controlled Study of Zileuton CR Tablets Versus Placebo in Adult Patients With Poorly Controlled Asthma Patients on Moderate Dose Inhaled Corticosteroids (ICS)
Brief Title: Zileuton CR vs Placebo in Poorly Controlled Asthma Patients on Moderate Dose ICS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slower than anticipated enrollment
Sponsor: Critical Therapeutics (Industry)
Responsible Party: Cornelis Wortel MD PhD/Acting CMO, Critical Therapeutics/Clinquest Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTI-03-C07-401
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Asthma
Keywords: Asthma; ICS; 5-LO Inhibition; Leukotrienes; Asthma control; Asthma exacerbations
MeSH Terms: conditions — Asthma | interventions — zileuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Zileuton CR
  Interventions: Drug: Zileuton CR
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zileuton CR — Zileuton CR tablets 2x600mg BID for 24 weeks
  Other Names: ZYFLO CR
  Arms: 1
Drug: Placebo — Placebo tablets 2x600mg BID for 24 weeks
  Arms: 2

SUMMARY:
Asthma is a chronic inflammatory disorder of the airways with a variety of inflammatory processes contributing to the pathogenesis. The inflammation leads to a state of increased airway responsiveness and reversible airway obstruction that causes the recurrent symptoms of asthma. Despite the variety of treatments available for asthma, none are curative, and the disease continues to place a burden on society in terms of morbidity, reduced quality of life (QOL), and ever increasing healthcare costs. The prevalence of asthma continues to increase with current data suggesting that since 1980, adult asthma cases have increased by 75% and in children under 5 years of age the prevalence has increased by 160%.1 Additionally, studies have suggested that the disease severity has been underestimated and that more patients may be classified as having moderate to severe persistent disease.2 Inhaled corticosteroids (ICS) have been the cornerstone of anti-inflammatory treatment for decades and have been shown to improve lung function, decrease symptoms, and reduce asthma exacerbations.3 However, many patients are still inadequately controlled despite treatment according to current asthma management guidelines and have a significant unmet medical need. Such patients are at high risk of serious exacerbations and asthma-related mortality.4 Combining long-acting β2-agonists (LABAs) with low dose ICS has been shown to improve asthma control over using higher doses of ICS alone. However, LABAs act mainly at the bottom of the inflammatory cascade and there are concerns that they may mask underlying inflammation.5 Recently, leukotriene receptor antagonists have been added to ICS as second-line therapy in the management of asthma. Zileuton has been extensively studied in inflammatory diseases such as asthma, in which leukotrienes mediate inflammation.

The aim of this study is to assess the effect of zileuton controlled-release (CR; 1200 mg 2-times daily [BID]) on pulmonary function, asthma control, and symptomatic response in adult patients with asthma poorly controlled on moderate dose ICS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 12-70 years of age (inclusive).
2. Diagnosis of asthma for at least 6 months.
3. Morning FEV1 of 40-80% normal.
4. Demonstrated reversible airflow restriction.
5. Non-smokers.
6. On moderate doses of ICS with inadequate asthma control.
7. Signed ICF

Exclusion Criteria:

1. Diagnosis of COPD.
2. Uncontrolled systemic illness.
3. Hypersensitivity to any component of ZYFLO CR
4. Any patient with an unscheduled visit to an ER or hospital for asthma exacerbation within past 3 months.
5. History of hepatitis or active liver disease.
6. ALT greater than 3xULN.
7. History of HIV infection
8. Recent history of drug or alcohol abuse.
9. Oral corticosteroids within one month, cromolyn sodium or nedocromil within 14 days, theophylline, LABA, ZYFLO, or leukotriene modifiers, warfarin or propranolol, inhaled anti-cholinergics, or combination LABA/ICS.
10. Omalizumab within 3 months.
11. Pregnant female.
12. Participation with 30 days in investigational study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-05 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function measures | 3 and 6 months

SECONDARY OUTCOMES:
Asthma exacerbations, ACQ, AQLQ, safety | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis Wortel, MD, PhD, Study Director — Critical Therapeutics/Clinquest Inc
Locations (1):
- Critical Therapeutics, Lexington, Massachusetts, United States

REFERENCES:
- See also: Specific Educational Information on Zileuton CR (Zyflo CR) — http://www.zyflocr.com